CLINICAL TRIAL: NCT06669026
Title: Therapeutic Efficacy of Local Vitamin D Drug as an Adjunct to Mechanical Debridement in the Treatment of Periodontitis
Brief Title: The Proposed Study Aims to Investigate the Impact of Adjunctive Vitamin D Gel Application on Gingival Crevicular Fluid Levels of Alkaline Phosphatase and Interleukin-8 in Periodontitis Patients Undergoing Phase 1 Periodontal Therapy. By Elucidating the Molecular Mechanisms Underlying the Therapeutic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: A0103023OM
Record Dates: First submitted 2024-10-23; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Intervention Model Description: Group 1: vitamin D3-loaded Poly lactic-co-glycolic acid (PLGA) nanoparticles gel as an adjunct to mechanical debridement.
  * Group 2: vitamin D3 gel (regular non-nanoparticle form) as an adjunct to mechanical debridement.
  * Group 3: placebo gel as an adjunct to mechanical debridement.
  * Group 4: only mechanical debridement.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- vitamin D3-loaded Poly lactic-co-glycolic acid nanoparticles gel adjunct to mechanical debridement (Experimental): vitamin D3-loaded Poly lactic-co-glycolic acid nanoparticles gel adjunct to mechanical debridement, and Interleukin 8/alkaline phosphatase Elisa analysis Frequency: once a week for 8 consecutive weeks Dosage, up to periodontal pocket fil
  Interventions: Dietary Supplement: vitamin D loaded Poly lactic-co-glycolic acid nanoparticles gel; Procedure: only mechanical debridement
- vitamin D3 gel (regular non-nanoparticle form) as an adjunct to mechanical debridement. (Active Comparator): vitamin D3 gel (regular non-nanoparticle form) as an adjunct to mechanical debridement, and Interleukin 8/alkaline phosphatase Elisa analysis Frequency: once a week for 8 consecutive weeks Dosage, up to periodontal pocket fil
  Interventions: Dietary Supplement: vitamin D3 gel (regular non-nanoparticle form); Procedure: only mechanical debridement
- Poly lactic-co-glycolic acid nanoparticles placebo gel adjunct to mechanical debridement. (Placebo Comparator): Poly lactic-co-glycolic acid nanoparticles placebo gel adjunct to mechanical debridement, and Interleukin 8/alkaline phosphatase Elisa analysis Frequency: once a week for 8 consecutive weeks Dosage, up to periodontal pocket fil
  Interventions: Other: Poly lactic-co-glycolic acid nanoparticles placebo gel; Procedure: only mechanical debridement
- only mechanical debridement only (Sham Comparator): only mechanical debridement only.
  Interventions: Procedure: only mechanical debridement
- Healthy patients (No Intervention): healthy patients, only added for Interleukin 8 and alkaline phosphatase Elisa analysis

INTERVENTIONS:
Dietary Supplement: vitamin D loaded Poly lactic-co-glycolic acid nanoparticles gel — Scaling and root debridement then inject gel in the pocket
  Arms: vitamin D3-loaded Poly lactic-co-glycolic acid nanoparticles gel adjunct to mechanical debridement
Dietary Supplement: vitamin D3 gel (regular non-nanoparticle form) — Scaling and root debridement then inject gel in the pocket
  Arms: vitamin D3 gel (regular non-nanoparticle form) as an adjunct to mechanical debridement.
Other: Poly lactic-co-glycolic acid nanoparticles placebo gel — Scaling and root debridement then inject gel in the pocket
  Arms: Poly lactic-co-glycolic acid nanoparticles placebo gel adjunct to mechanical debridement.
Procedure: only mechanical debridement — Scaling and root debridement
  Arms: Poly lactic-co-glycolic acid nanoparticles placebo gel adjunct to mechanical debridement.; only mechanical debridement only; vitamin D3 gel (regular non-nanoparticle form) as an adjunct to mechanical debridement.; vitamin D3-loaded Poly lactic-co-glycolic acid nanoparticles gel adjunct to mechanical debridement

SUMMARY:
The proposed study aims to investigate the impact of adjunctive vitamin D gel application on gingival crevicular fluid levels of alkaline phosphatase and interleukin-8 in periodontitis patients undergoing phase 1 periodontal therapy. By elucidating the molecular mechanisms underlying the therapeutic effects of vitamin D, this research seeks to contribute to the development of more effective treatment strategies for periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with attachment loss 3-4 mm
* periodontal pocket ≤ 5 mm

Exclusion Criteria:

* - Patients with sensitivity to the medication used in the study.
* Patients with a history of antibiotic use or anti-inflammatory drugs during the previous 3 months prior to the study.
* Patients with systemic diseases.
* Pregnant and lactating females.
* Smokers and tobacco chewers.
* Patients not compliant with oral hygiene procedures.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Periodontal Assessment | 12 weeks
  Periodontal Index

SECONDARY OUTCOMES:
Interleukin 8 | 8 weeks
  level of interleukin 8 in gingival crevicular fluid will be tested via elisa
alkaline phosphatase | 8 weeks
  level of alkaline phosphatase in gingival crevicular fluid will be tested via elisa

CONTACTS AND LOCATIONS:
Locations (1):
- Alaaeldin Ahmed Taha, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided